CLINICAL TRIAL: NCT06540313
Title: Efficacy, Safety and Neural Mechanism of Stellate Ganglion Block in the Treatment of Anxiety.
Brief Title: Efficacy, Safety and Neural Mechanism of Stellate Ganglion Block in the Treatment of Anxiety. Disorder.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, associate professor, Nanjing Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SGB-KY-2024
Record Dates: First submitted 2024-07-09; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorders; Stellate Ganglion Block
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Relieve anxiety symptoms (Experimental)
  Interventions: Other: Stellate Ganglion Block
- Restore mental function (Experimental)
  Interventions: Other: Stellate Ganglion Block
- Verify Stellate Ganglion Block security (Experimental)
  Interventions: Other: Stellate Ganglion Block
- Explore the Stellate Ganglion Block intervention mechanism (Experimental)
  Interventions: Other: Stellate Ganglion Block

INTERVENTIONS:
Other: Stellate Ganglion Block — Stellate ganglion block refers to the injection of local anesthetic drugs into tissues around and near SG to regulate the tension of the sympathetic nervous system, inhibit the outflow of the sympathetic nerve in the innervation area of the stellate ganglion to the ipsilateral head, neck, chest and upper limb, and finally achieve the role of regulating the autonomic nervous system, circulatory system, endocrine system and immune system of the human body to maintain dynamic balance. It is used to treat a variety of pain and non-pain diseases.

SUMMARY:
1. In this study, ultrasound-guided Stellate Ganglion Block(SGB) will be used in the treatment of anxiety disorders, combined with relevant scales, HRV indicators and resting state functional magnetic resonance data, to explore the safety and effectiveness of SGB in the treatment of anxiety disorders, and to explore whether its mechanism of action is related to the excitability of sympathetic nervous system and the activity changes of insular cortex.
2. Verify the following hypothesis:

(1) SGB is a safe, well-tolerated and acceptable treatment technique; (2) After SGB treatment, the anxiety symptoms of the patients were relieved to a certain extent and the psychological function was restored; (3) The sympathetic excitability of patients after SGB treatment is reduced, and this effect can be monitored by heart rate variability; (4) The activity of insular cortex decreased after SGB treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years old
2. Diagnosed with various types of anxiety disorders according to the DSM-5, and meet the diagnostic criteria for pain disorders
3. Right-handed
4. Voluntarily join the study and sign the informed consent.

Exclusion Criteria:

1. Suicidal thoughts and behaviors
2. serious physical disease
3. diseases of the nervous system or other mental diseases
4. Contraindications for MRI examination
5. During pregnancy or lactation
6. Allergy to narcotic drugs
7. Contraindications with stellate ganglion block

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability index | 8 weeks
  Heart rate variability is an important index to measure the tone and balance of the sympathetic and parasympathetic nerves. Heart rate variability can reflect the sympathomympathetic nerve function of patients with anxiety disorder.
Insular cortex activity | 8 weeks
  The insular cortex is the most important cortical region that controls sympathetic and parasympathetic mediated cardiovascular regulation and plays a key role in maintaining body homeostasis. However, a recent study found that the change of heart rate in mice can affect anxiety symptoms through the insular cortex, so it is speculated that SGB may induce the change of insular cortex activity by regulating the activity of sympathetic nervous system, thus alleviating anxiety symptoms.
Numeric Rating Scale | 8 weeks
  In this study, Numeric Rating Scale was used to explore the efficacy of stellate ganglion block in the treatment of anxiety disorders. The scale consists of 11 numbers from 0 to 10. Patients use 11 numbers, from 0 to 10, to describe the intensity of the pain, and the higher the number, the worse the pain. 0 means no pain, 1 to 3 means mild pain (pain does not affect sleep), 4 to 6 means moderate pain, 7 to 9 means severe pain (can not fall asleep or wake up in sleep), and 10 means severe pain.
Hamilton Anxiety Rating Scale | 8 weeks
  In this study, Hamilton Anxiety Rating Scale was used to explore the efficacy of stellate ganglion block in the treatment of anxiety disorders.There are 14 items in the scale, and all items are scored with a 5-level scoring method ranging from 0 to 4 points. The sum of the scores of each item is the total score of the scale. A total score of <7 indicates no anxiety symptoms, a score of 7-13 indicates possible anxiety symptoms, a score of 14-20 indicates certain anxiety symptoms, a score of 21-28 indicates obvious anxiety symptoms, and a score of ≥29 indicates possible severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No